CLINICAL TRIAL: NCT02081300
Title: Phase 3, Active-Controlled, Safety and Efficacy Trial of Oral Testosterone Undecanoate (TU, LPCN 1021) in Hypogonadal Men
Brief Title: Safety and Efficacy of Oral LPCN 1021 in Men With Low Testosterone or Hypogonadism
Acronym: SOAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lipocine Inc. (Industry)
Collaborators: Syneos Health (Other); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPCN 1021-13-001
Record Dates: First submitted 2014-02-20; First posted 2014-03-07 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Male Hypogonadism
Keywords: Testosterone; Male hypogonadism; Low testosterone; LPCN 1021; Androgel; Testim; Testopel; Fortesta; Axiron.; Hypogonadism; Eunuchism; Gonadal Disorders; Endocrine System Diseases; Testosterone enanthate; Testosterone undecanoate; Testosterone 17 beta-cypionate; Methyltestosterone; Androgens; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Physiological Effects of Drugs; Pharmacologic Actions; Antineoplastic Agents, Hormonal; Antineoplastic Agents; Anabolic Agents
MeSH Terms: conditions — Eunuchism; Hypogonadism; Gonadal Disorders; Endocrine System Diseases | interventions — testosterone undecanoate; Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral testosterone undecanoate, LPCN 1021 (Experimental): Oral testosterone undecanoate: Initial dose: 225 mg TU BID. Dose titrated up to 300 mg TU BID or down to 150 mg TU BID based on serum T at Week 3 and 7.
  Interventions: Drug: Oral testosterone undecanoate, LPCN 1021
- Topical testosterone gel 1.62 % (Other): Topical testosterone gel 1.62%: Initial dose: 40.5 mg T once daily. Dose titrated down to 20.25 mg or up to 81 mg based on serum T on Days 14 and 28
  Interventions: Drug: Topical testosterone gel 1.62 %

INTERVENTIONS:
Drug: Oral testosterone undecanoate, LPCN 1021
  Arms: Oral testosterone undecanoate, LPCN 1021
Drug: Topical testosterone gel 1.62 %
  Arms: Topical testosterone gel 1.62 %

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an oral testosterone undecanoate formulation for use as testosterone-replacement therapy in men with low testosterone.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of primary hypogonadism (congenital or acquired) or hypogonadotropic hypogonadism (congenital or acquired).
2. Serum total testosterone < 300 ng/dL based on 2 consecutive blood samples

Exclusion Criteria:

A subject will not be eligible for study participation if he meets any of the following criteria.

1. History of significant sensitivity or allergy to androgens, castor oil or product excipients.
2. Clinically significant findings in the prestudy examinations.
3. Abnormal prostate digital rectal examination (DRE) with palpable nodule(s) or I-PSS score > 19 points.
4. Body mass index (BMI) ≥ 38 kg/m2.
5. Clinically significant abnormal laboratory values
6. Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus antibodies (HIV Ab).
7. History of seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
8. History of gastric surgery, cholecystectomy, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
9. History of any clinically significant illness, infection, or surgical procedure within 1 month prior to study drug administration.
10. History of stroke or myocardial infarction within the past 5 years.
11. History of, or current or suspected, prostate or breast cancer.
12. History of diagnosed, severe, untreated, obstructive sleep apnea.
13. History of abuse of alcohol or any drug substance in the opinion of the investigator within the previous 2 years.
14. History of long QT syndrome or unexplained sudden death in a first degree relative (parent, sibling, or child).
15. Concurrent treatment with medications which may impact the absorption, distribution, metabolism or excretion of testosterone undecanoate (TU) or place the subject at risk for treatment with testosterone.
16. Subject has a partner who is currently pregnant or planning pregnancy during the course of the clinical trial.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Proportion of LPCN 1021-treated subjects who achieve a total testosterone concentration [Cavg] between 300 - 1140 ng/dL. | Following 13 weeks of treatment

SECONDARY OUTCOMES:
Percentage of LPCN 1021-treated subjects with maximum serum T concentrations (Cmax) values that are (a) less than 1500 ng/dL; (b) between 1800 and 2500 ng/dL, and (c) greater than 2500 ng/dL | Following 13 weeks of treatment
Change from baseline in patient reported outcomes for LPCN 1021 (i.e., International Prostate Symptom Score [I-PSS], Psychosexual Daily Questionnaire [PDQ], Short Form-36 Questionnaire [SF-36]) | 52 weeks
Change from baseline to 52 weeks in safety laboratory parameters (i.e., clinical chemistry, hematology, PSA) | 52 weeks
Number of subjects with adverse events during 52 weeks of treatment | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DelConte, MD, Study Director — Chief Medical Director, Lipocine, Inc.